CLINICAL TRIAL: NCT04109976
Title: A Multicenter, Randomized, Open-Label Study to Evaluate the Safe and Effective Use of the Prefilled Safety Syringe or Auto-Injector for the Subcutaneous Self-Injection of Bimekizumab Solution by Subjects With Active Psoriatic Arthritis
Brief Title: A Study to Evaluate the Safe and Effective Use of the Prefilled Safety Syringe or the Auto-injector for the Subcutaneous Self-injection of Bimekizumab Solution by Subjects With Active Psoriatic Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DV0004; 2018-004725-86 (EudraCT Number)
Record Dates: First submitted 2019-09-27; First posted 2019-10-01 (Actual); Results first posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic Arthritis; PsA; Auto-Injector; Bimekizumab
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — bimekizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bimekizumab-SS (Experimental): Study participants randomized to this arm will receive assigned bimekizumab dose regimen using the prefilled safety syringe (SS).
  Interventions: Drug: Bimekizumab
- Bimekizumab-AI (Experimental): Study participants randomized to this arm will receive assigned bimekizumab dose regimen using the auto-injector (AI).
  Interventions: Drug: Bimekizumab

INTERVENTIONS:
Drug: Bimekizumab — Study participants will receive bimekizumab at pre-specified time points.
  Other Names: UCB4940; BKZ

SUMMARY:
The purpose of the study is to evaluate for each self-injecting device presentation the ability of subjects with psoriatic arthritis (PsA) to safely and effectively self-inject bimekizumab at study start and 4 weeks after training in self-injection technique using the bimekizumab safety syringe (SS) or the bimekizumab auto-injector (AI).

ELIGIBILITY:
Inclusion Criteria:

* Subject fulfills all inclusion criteria for the PA0012 [NCT04009499] study
* Subject is considered reliable and capable of adhering to the DV0004 protocol (eg, able to understand and complete questionnaires, able to use investigational self-injecting device presentations according to the instructions for use (IFU), and able to adhere to the visit schedule) according to the judgment of the Investigator
* Subject is willing to self-inject

Exclusion Criteria:

-Subjects are not permitted to enroll in DV0004 if any of the PA0012 [NCT04009499] study exclusion criteria are met

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2020-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (47):
- United States (20):
  - Dv0004 50024, Boise, Idaho
  - Dv0004 50028, Lexington, Kentucky
  - Dv0004 50023, Baton Rouge, Louisiana
  - Dv0004 50015, Hagerstown, Maryland
  - Dv0004 50026, Wheaton, Maryland
  - Dv0004 50019, Lansing, Michigan
  - Dv0004 50016, St Louis, Missouri
  - Dv0004 50005, Freehold, New Jersey
  - Dv0004 50029, Albuquerque, New Mexico
  - Dv0004 50010, Brooklyn, New York
  - Dv0004 50125, Charlotte, North Carolina
  - Dv0004 50031, Salisbury, North Carolina
  - Dv0004 50040, Dayton, Ohio
  - Dv0004 50020, Duncansville, Pennsylvania
  - Dv0004 50006, Wyomissing, Pennsylvania
  - Dv0004 50008, Johnston, Rhode Island
  - Dv0004 50001, Jackson, Tennessee
  - Dv0004 50036, Mesquite, Texas
  - Dv0004 50009, Waco, Texas
  - Dv0004 50050, Beckley, West Virginia
- Czechia (6):
  - Dv0004 40061, Brno
  - Dv0004 40009, Pardubice
  - Dv0004 40063, Prague
  - Dv0004 40066, Prague
  - Dv0004 40010, Uherské Hradiště
  - Dv0004 40012, Zlín
- Dv0004 40029, Hamburg, Germany
- Dv0004 40079, Szentes, Hungary
- Poland (14):
  - Dv0004 40038, Elblag
  - Dv0004 40088, Elblag
  - Dv0004 40096, Gdynia
  - Dv0004 40042, Krakow
  - Dv0004 40092, Krakow
  - Dv0004 40037, Lublin
  - Dv0004 40091, Nowa Sól
  - Dv0004 40044, Poznan
  - Dv0004 40118, Torun
  - Dv0004 40041, Warsaw
  - Dv0004 40097, Warsaw
  - Dv0004 40098, Warsaw
  - Dv0004 40039, Wroclaw
  - Dv0004 40043, Wroclaw
- Russia (5):
  - Dv0004 20005, Moscow
  - Dv0004 20013, Petrozavodsk
  - Dv0004 20004, Saint Petersburg
  - Dv0004 20014, Ulyanovsk
  - Dv0004 20015, Yaroslavl

IPD SHARING:
Plan to Share IPD: Yes
Data from this study may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.clinicalstudydatarequest.com and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal. This plan may change if a determination is made that the data cannot be adequately anonymized.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this study may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.clinicalstudydatarequest.com and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- See also: Product Information — https://www.ema.europa.eu/en/documents/product-information/bimzelx-epar-product-information_en.pdf
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll study participants in Aug 2019 and concluded in Nov 2020. This study is a substudy to PA0012 (NCT04009499).
Pre-assignment Details: Participant Flow refers to the Enrolled Set.
Groups:
- BKZ-SS-1mL 160 mg Q4W: Participants self-injected bimekizumab (BKZ) 160 milligrams (mg) solution every 4 weeks (Q4W) as a subcutaneous (sc) injection with bimekizumab-Safety Syringe-1 milliliter (mL) (BKZ-SS-1mL) device presentation (ie. 2 self-injections) at Baseline and at Week 4.
- BKZ-AI-1mL 160 mg Q4W: Participants self-injected BKZ 160 mg solution Q4W as a sc injection with bimekizumab-Auto-Injector-1mL (BKZ-AI-1mL) device presentation (ie. 2 self-injections) at Baseline and at Week 4.
Period: Overall Study
Arm/Group | BKZ-SS-1mL 160 mg Q4W | BKZ-AI-1mL 160 mg Q4W
Started | 107 | 107
Completed | 106 | 107
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set (SS) consisted of all study participants who received at least 1 dose of bimekizumab by the indicated self-injection investigational device presentation (bimekizumab-SS-1mL [SS-s] and bimekizumab-AI-1mL [SS-a]).
Groups:
- BKZ-SS-1mL 160 mg Q4W: Participants self-injected BKZ 160 mg solution Q4W as a sc injection with BKZ-SS-1mL device presentation (ie. 2 self-injections) at Baseline and at Week 4.
- BKZ-AI-1mL 160 mg Q4W: Participants self-injected BKZ 160 mg solution Q4W as a sc injection with BKZ-AI-1mL device presentation (ie. 2 self-injections) at Baseline and at Week 4.
- Total: Total of all reporting groups
Arm/Group | BKZ-SS-1mL 160 mg Q4W | BKZ-AI-1mL 160 mg Q4W | Total
Number analyzed (Participants) | 107 | 107 | 214
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 94 | 91 | 185
  >=65 years | 13 | 16 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.3 (13.2) | 51.5 (11.9) | 49.9 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 54 | 108
  Male | 53 | 53 | 106
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 106 | 107 | 213
  Other/Mixed | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 106 | 107 | 213
  Hispanic or Latino | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Able to Self-administer Safe and Effective Injections Using the Bimekizumab Safety Syringe (BKZ-SS) or the Bimekizumab Auto-injector (BKZ-AI) at Week 4
Description: Safe and effective self-injection was evaluated by the study personnel and was defined as: - Complete dose delivery: Participant self-injected the complete dose of bimekizumab as confirmed by a visual inspection of the bimekizumab-safety syringe (SS) or the bimekizumab-auto-injector (AI) which shows that the investigational medicinal product (IMP) was delivered completely (ie, container is empty), and - No Adverse Device Effects (ADEs) that would preclude continued use of the device for self-injection (ie, no serious ADEs (SADEs) and/or ADEs leading to withdrawal).
Time Frame: Week 4
Population: The Full Analysis Set for device presentation bimekizumab-SS-1mL (FAS-s) and bimekizumab-AI-1mL (FAS-a) consisted of all study participants in the SS-s and SS-a who self-injected at least 1 dose of bimekizumab using the given device presentation and who had an assessment of self-injection. Here, Number of Participants analyzed signifies participants who were evaluable for the assessment.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | BKZ-SS-1mL 160 mg Q4W | BKZ-AI-1mL 160 mg Q4W
Number analyzed (Participants) | 105 | 104
percentage of participants | 100 [97.2 to 100] | 100 [97.2 to 100]

2. Secondary Outcome: Percentage of Participants Able to Self-administer Safe and Effective Injections Using the Bimekizumab Safety Syringe (BKZ-SS) or the Bimekizumab Auto-injector (BKZ-AI) at Baseline
Description: Safe and effective self-injection was evaluated by the study personnel and was defined as: - Complete dose delivery: Participant self-injected the complete dose of bimekizumab as confirmed by a visual inspection of the bimekizumab-SS or the bimekizumab-AI which shows that the IMP is delivered completely (ie, container is empty), and - No ADEs that would preclude continued use of the device for self-injection (ie, no SADEs and/or ADEs leading to withdrawal).
Time Frame: Baseline
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | BKZ-SS-1mL 160 mg Q4W | BKZ-AI-1mL 160 mg Q4W
Number analyzed (Participants) | 106 | 106
percentage of participants | 100 [97.2 to 100] | 100 [97.2 to 100]

ADVERSE EVENTS:
Time Frame: From Baseline up to Week 5
Description: Treatment emergent adverse device events (TEADEs) were defined as adverse event related to study device that have a start date on or following the first self-administration of study treatment through the final self-administration of study treatment plus 7 days. As Pre-specified in SAP, only those AEs related to the use of the investigational medical devices BKZ-SS or BKZ-AI (based on the Investigator's judgment) were assessed and have been reported in this section.
Arm/Group | BKZ-SS-1mL 160 mg Q4W | BKZ-AI-1mL 160 mg Q4W
All-Cause Mortality (participants affected / at risk) | 0/107 | 0/107
Serious Adverse Events (participants affected / at risk) | 0/107 | 0/107
Other Adverse Events (participants affected / at risk) | 0/107 | 0/107

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/76/NCT04109976/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/76/NCT04109976/SAP_001.pdf